CLINICAL TRIAL: NCT05053490
Title: Static Versus Dynamic Stretching; Short Term Effects On Physical Performance In Non-Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01012 Arooba.
Record Dates: First submitted 2021-08-12; First posted 2021-09-22 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Physical Fitness
Keywords: Static and dynamic stretching
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants of group A will perform static stretches and group B will perform dynamic stretching. After a gap of 3 days, interventions will be switched, now group A will perform dynamic stretching and group B will perform static stretching.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Stretching (Experimental): Participants will perform static stretching on day 1 and dynamic stretching after the switching.
  Interventions: Other: Static Stretching
- dynamic stretching (Experimental): Participants will perform dynamic stretching on day 1 and static stretching after the switching.
  Interventions: Other: dynamic stretching

INTERVENTIONS:
Other: Static Stretching — Static stretches are those in which you stand, sit or lie still and hold a single position for a period of time.
  Arms: Static Stretching
Other: dynamic stretching — Dynamic stretching involves making active movements that stretch the muscles to their full range of motion.
  Arms: dynamic stretching

SUMMARY:
This study will compare the short-term effects of static and dynamic stretching on the physical performance of undergraduate students who are not involved in athletic activities. It will be observed if a significant difference lies between these stretchings.

DETAILED DESCRIPTION:
The individual participant will be assessed at baseline and then stretching will be performed after that. Group A will perform static stretching and group B will perform dynamic stretching. Immediate assessment will be done after 5 minutes, a second assessment will be done after 6 hours and a third one will be done after 24 hours to measure the short-term effects.

After that, a gap of 3 days will be given and stretching will be performed again. Now, group A will perform dynamic stretching and group B will perform static stretching. A similar assessment will be repeated after 5 minutes then 6 hours and then after 24 hours to determine the difference.

ELIGIBILITY:
Inclusion Criteria:

* Male undergraduate students aged between 18-25
* Lower Limb range; Hip SLR>80 degree Knee flexion >130 degree Ankle dorsiflexion >20 degree
* Those who fall under normal BMI range

Exclusion Criteria:

* acute injuries of the lower limb.
* active participants of sports and any training programs.
* lower limb disabilities.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males were selected because girls could not perform outdoor physical performance tests because of cultural issues.
Enrollment: 54 (Estimated)
Dates: Start 2021-12-24 (Estimated); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Endurance in meters. | 5 minutes
  Cooper 12-minute walk/run test for endurance.
Vertical jump in inches. | 5 minutes
  Vertical Jump Test (Sargent Jump, Vertical Leap) for strength.
Agility in seconds. | 5 minutes.
  Modified Illinois Agility Test for agility.
Flexibility in inches. | 5 minutes
  Sit-and-reach test for flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No